CLINICAL TRIAL: NCT06579781
Title: Rigorous Evaluation of Morehouse School of Medicine's Parent Toolkit 2.0 Intervention (Morehouse Family Health Study)
Brief Title: Evaluation of Parent Toolkit 2.0 (Morehouse Family Health Study)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Child Trends (Other)
Responsible Party: Principal Investigator, Jennifer Manlove, Principal Investigator, Child Trends
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Child Trends
Record Dates: First submitted 2024-08-20; First posted 2024-08-30 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2024-10

CONDITIONS: Sexual Behavior; Adolescent Behavior; Sexually Transmitted Diseases; Contraception Behavior; Parent-Child Relations
Keywords: teen pregnancy; STIs; parent-teen communication; parenting; adolescent sexual health
MeSH Terms: conditions — Sexual Behavior; Adolescent Behavior; Sexually Transmitted Diseases; Contraception Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Condition (Active Comparator): Adult participants in the control condition will receive access to an online general health guide for parents that was adapted for this study from a pre-existing health guide.
  Interventions: Behavioral: Morehouse Family Health Study's General Health Guide
- Treatment Condition (Experimental): Adult participants in the treatment condition will receive access to the Parent Toolkit 2.0 intervention, which includes an online interactive guide, four videos modeling parent-teen communication around sex and contraception, and two group-based, virtual sessions with other parents and caregivers.
  Interventions: Behavioral: Morehouse Family Health Study's Parent Toolkit 2.0

INTERVENTIONS:
Behavioral: Morehouse Family Health Study's Parent Toolkit 2.0 — Parent Toolkit 2.0 is designed to equip parents and caregivers with skills to talk to their teens about sex and contraception and ultimately influence their teens' decision-making and behaviors around sex. The Georgia Campaign for Adolescent Power & Potential (GCAPP) developed the Parent Toolkit intervention. Morehouse School of Medicine's (MSM) Health Promotion Research Center tested and adapted it through an OPA Innovation Network grant, creating Parent Toolkit 2.0.
  Arms: Treatment Condition
Behavioral: Morehouse Family Health Study's General Health Guide — General Health Guide provides information to parents on how to promote health in their families.
  Arms: Control Condition

SUMMARY:
Child Trends will conduct a randomized control trial evaluation of Parent Toolkit 2.0, an innovative intervention for parents and caregivers of middle and high school students. Child Trends will collaborate with Morehouse School of Medicine and Tressa Tucker & Associates, LLC to implement and evaluate the program with 1,000 parent-teen pairs across Georgia. The program includes three components that will be delivered across a three-week period: (1) an online self-paced Parent Guide with information, tips, tools, and resources on adolescent health, including sexual health; (2) four videos modeling parent-teen communication around sex and contraception; and (3) two group-based sessions for parent participants to discuss program content and improve communication skills. The program aims to increase parent knowledge and parent-teen communication about adolescent health, sexual health, and relationships to help youth adopt health-promoting behaviors such as delaying sexual initiation and increasing contraceptive use.

DETAILED DESCRIPTION:
Child Trends, in partnership with the Morehouse School of Medicine (MSM), will implement Parent Toolkit 2.0. The Georgia Campaign for Adolescent Power & Potential developed the Parent Toolkit intervention and Morehouse School of Medicine's (MSM) Health Promotion Research Center tested and adapted it through an OPA Innovation Network grant.

Child Trends plans to conduct an individual randomized controlled trial (RCT) to evaluate the effectiveness of Parent Toolkit 2.0 in delaying sexual initiation and increasing contraceptive use among youth who engage in sexual activity. Youth outcomes are expected to improve as a result of the expansion of parental knowledge and improvement of parent-teen communication about adolescent health, sexual health, and relationships. Associated outcomes will be measured through two surveys, one of which will be distributed immediately after the intervention ends while the other will be administered nine months after the end of the intervention.

The intended population is youth ages 12-15 living in rural and micropolitan areas in central, north, and southeast Georgia, and their parents or caregivers. A "caregiver" in this context is defined as someone who lives with the child at least 50 percent of the time and who is one of the main people responsible for the child. The parents or caregivers will be the program participants since they are the intended recipients of all intervention-related resources such as the toolkit, videos, and group-based virtual sessions. By contrast, the youth enrolled in the study will not directly engage in the programming.

As a part of this study, treatment group parent/caregiver participants will be asked to:

* Review a self-paced parent guide and four videos modeling parent-teen communication on Canvas
* Attend two 1-hour group sessions with other parents
* Complete baseline and post-intervention surveys
* Participate in an optional focus group discussion

Control group parent/caregiver participants will be asked to:

* Review a self-paced parent guide on Canvas
* Complete baseline and post-intervention surveys
* Participate in an optional focus group discussion

Treatment and control group youth participants will be asked to:

* Complete baseline, post-intervention, and nine-month follow-up surveys
* Participate in an optional focus group discussion

ELIGIBILITY:
Inclusion Criteria for Adult Participants:

* 25 to 70 years old
* Lives in an eligible zip code in Georgia
* Parent or caregiver of 12- to 15-year-old child who wants to participate in this study with them
* Lives with child at least 50% of the time

Exclusion Criteria for Adult Participants:

* Lives in a home with a child who is already enrolled in this study
* Raises child with an adult who is already enrolled in this study

Inclusion Criteria for Child Participants:

* 12-15 years old
* Lives with a parent or caregiver who wants to participate in this study with them
* Able to complete surveys on own or with help of support person

Exclusion Criteria for Child Participants:

- Does not have their own email address or phone number

Ages: 12 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2000 (Estimated)
Dates: Start 2024-10-21 (Actual); Primary Completion 2028-04-30 (Estimated); Study Completion 2028-09-29 (Estimated)

PRIMARY OUTCOMES:
No recent penile-vaginal or oral sex | 9 months after end of program
  Yes = Has not had penile-vaginal or oral sex in past 3 months; No = Has had penile-vaginal or oral sex in past three months.

SECONDARY OUTCOMES:
No recent penile-vaginal sex | 9 months after end of program
  Yes = Has not had consensual penile-vaginal sex in past 3 months; No = Has had consensual penile-vaginal sex in past 3 months.
Never had penile-vaginal sex | 9 months after end of program
  Yes = Has never had consensual penile-vaginal sex; No = Has had consensual penile-vaginal sex.
Never had penile-vaginal or oral sex | 9 months after end of program
  Yes = Has never had consensual penile-vaginal or oral sex; No = Has had consensual penile-vaginal or oral sex.
Protected penile-vaginal sex or no penile-vaginal sex | 9 months after end of program
  Yes = Always used pill, shot, patch, ring, IUD, implant, or condom during penile-vaginal sex OR did not have penile-vaginal sex; No = Had penile-vaginal sex without using pill, shot, patch, ring, IUD, implant, or condom every time
Parent-child communication | Immediately after end of program and 9 months after end of program
  Score of talking with parent/caregiver about important topics, such as online safety, love languages, healthy relationships, peer pressure and bullying, puberty, sexual activity, reproduction, birth control, condoms, STIs, and going to the doctor for sexual health care. Scores will range from 0 to 16, with a higher score indicating a better outcome.
Parent-child relationship closeness | Immediately after end of program and 9 months after end of program
  Score of parent-child relationship, including frequency of having fun doing something with parent, having a good conversation with parent about something that matters to the youth, going to parent when the youth was feeling unhappy or needing help, resolving conflicts together with parent, and comfort talking with parent about important topics. Scores will range from 0 to 6, with a higher score indicating a better outcome.
Self-efficacy to avoid sex and to use contraceptives | Immediately after end of program and 9 months after end of program
  Score of confidence in being able to not have penis-in-vagina sex if the youth does not want to and to use birth control every time youth has penile-vaginal sex. Scores will range from 0 to 6, with higher scores indicating more self-efficacy.
Emotional wellbeing | Immediately after end of program and 9 months after end of program
  Score of mental health during past week, including feeling depressed or very sad, fearful, bothered by things that do not usually bother youth, trouble keeping mind on what youth is doing, that everything youth did used up a lot of their energy, hopeful about the future, hard to go to sleep or stay asleep, happy, lonely, could not get going. Scores will range from 0 to 30, with higher scores indicating better mental health.
Intention to avoid sex and to use contraceptives | Immediately after end of program and 9 months after end of program
  Score of intentions to not have penis-in-vagina sex in the next year and to use (or support their partner in using) birth control during penile-vaginal sex in next year. Scores will range from 0 to 3, with higher scores indicating stronger intentions.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Manlove, PhD, Principal Investigator — Child Trends
Locations (1):
- Community Outreach, Cairo, Georgia, United States

IPD SHARING:
Plan to Share IPD: No